CLINICAL TRIAL: NCT03997942
Title: The Effect of Proprioceptive Neuromuscular Facilitation and Mirror Therapy on Range of Motion, Pain, Functionality, Kinesophobia and Quality of Life in Patients With Upper Extremity Burns
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mine Seyyah, Msc Physiotherapist, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: Kartal Wound and Burn Center
Record Dates: First submitted 2019-06-18; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Burn; Arm
Keywords: burn, physiotherapy
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- proprioceptive neuromuscular facilitation: PNF will be applied to randomly selected patients.
  Interventions: Other: Effect of exercise
- Mirror therapy: Mirror therapy will be applied to randomly selected patients.
  Interventions: Other: Effect of exercise
- Standart therapy: Standard treatment will be applied to randomly selected patients.
  Interventions: Other: Effect of exercise

INTERVENTIONS:
Other: Effect of exercise — Once the data are available, we hope to have information about which of the exercise practices included in the rehabilitation program of acute upper extremity burn patients is more effective.

SUMMARY:
Purpose of the study; The aim of this study was to investigate the effect of two different exercise programs on joint patency, pain, functionality, kinesophobia and quality of life in upper extremity burn patients. Lütfi Kırdar Training and Research Hospital Burn and Wound Center and unilateral upper extremity burns will consist of individuals aged 18-65 years. 48 burn patients who volunteered to participate in the study will be included in the study. Demographic information of the cases will be recorded. Joint range of motion and pain will be evaluated with the Visual Analogue Scale (VAS) before and after the treatment program. Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire will be used to evaluate upper extremity functions. TAMPA Kinezophobia questionnaire will also be used for kinesiophobia. To evaluate the quality of life, Burn-Specific Health Scale developed for burn patients will be used.

DETAILED DESCRIPTION:
Joint range of motion of the subjects will be measured with a goniometer. Pain will be evaluated with the Visual Analogue Scale (VAS). In order to evaluate the upper extremity functions, the validity and reliability of the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire, conducted by Tülin Düger et al. The TAMPA Kinezophobia questionnaire, which has been validated and validated in 2011, will be used for kinesiophobia. The Burn-Specific Health Scale developed for burn patients will be used to evaluate the quality of life. The validity and reliability study of the questionnaire was conducted by Mehmet Adam et al.

ELIGIBILITY:
Inclusion Criteria: -18-65 years of age, -the unilateral upper extremity burn, -the understanding of the given information, the application of mirror therapy and the ability to accurately express the level of pain that prevents cognitive, affective and verbal communication There is no problem and no visual impairment, - Turkish reading and writing, - Paralysis, plaster, etc. that will prevent movement in the extremity opposite the burned extremity. to be cognitive enough to understand the surveys,

- Agreeing to participate voluntarily in the study -

Exclusion Criteria:

* T.C. Ministry of Health Kartal Lütfi Kırdar Training and Research Hospital Burn and Wound Center treated patients between the ages of 0-18,
* Burn patients who refused to participate in the study, - Patients with bilateral upper extremity burns

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Burn Patients
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-09-20 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Demographic information | 10 minutes
  Demographic information of the cases will be recorded.Age, cause of burn, burn zone, burn percentage will be recorded.
Joint range of motion | 15 minutes
  The goniometer will measure the range of motion.
Pain assesment | 5 minutes
  Pain will be assessed by visual pain scale.
Functional assesment | 15 minutes
  Shoulder-Arm Function Questionnaire will be used to evaluate upper extremity functions.
Fear of Motion | 10 minutes
  The Tampa Kinesophobia Questionnaire will be used to assess fear of movement.
Quality of Life Assesment | 15 minutes
  A scale specific to burn patients will be used to evaluate the quality of life.(Burn Specific Health Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Mine Seyyah, Study Chair — DrLutfiKirdar
Locations (1):
- Wound and Burn Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No